CLINICAL TRIAL: NCT01016223
Title: A Randomized Double Blind Placebo Controlled Study of the Effect of Swallowed Beclomethasone Dipropionate on Inflammatory Markers in Adult Patients With Eosinophilic Esophagitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Gisoo Ghaffari, Assistant professor of Medicine, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 32508
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Eosinophilic Esophagitis
Keywords: Eosinophilic esophagitis; Beclomethasone; Ultrasensitive CRP
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Beclomethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Beclomethasone dipropionate inhaler (Active Comparator)
  Interventions: Drug: Beclomethasone dipropionate
- Matched inhaler (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Beclomethasone dipropionate — Beclomethasone dipropionate 80 mcg two puffs twice daily for 8 weeks
  Arms: Beclomethasone dipropionate inhaler
Drug: placebo — Matched placebo swallowed two puffs twice daily
  Arms: Matched inhaler

SUMMARY:
The investigators hypothesize that swallowed beclomethasone leads not only to improvement of symptoms and decreased number of eosinophils in esophageal mucosa, but also to a decrease in other markers of tissue inflammation like mast cells, CD4+ T lymphocytes, IL4, IL-5, IL13, GM-CSF and TGF-beta as well as serum ultra-sensitive C-Reactive Protein (CRP). The investigators aim to characterize the response of esophageal inflammation to swallowed topical glucocorticoids, and identify biomarkers to assess response to treatment.

This research will elucidate the effect of treatment with beclomethasone on various inflammatory markers in EoE, which is currently not well-understood. This work will explore the pathophysiology of EoE, and has the potential to find a non-invasive biomarker such as high-sensitivity CRP that can be used to monitor the response to treatment.

DETAILED DESCRIPTION:
EoE is an increasingly recognized clinicopathological diagnosis, characterized by a marked accumulation of eosinophils in the esophageal mucosa.The presence of eosinophils and association of the disease with food allergy and allergic rhinitis suggests an atopic disease. Allergic diseases are associated with T-helper 2 lymphocytes (TH2) predominant cytokines such as interleukins 4, 5, 13 (IL4, IL5, IL13), which are known to induce IgE synthesis and promote eosinophilic infiltration. Granulocyte-Monocyte Colony Stimulating Factor (GM-CSF) and Transforming Growth Factor (TGF) - beta are cytokines which are associated with many eosinophilic disorders. Swallowed steroid is a conventional treatment that has been shown to improve symptoms and decrease number of eosinophils in the esophagus in patients with EoE. However, no studies have investigated the effect of swallowed steroid on markers of TH2 inflammation in adult patients with EoE.Currently repeated endoscopic biopsy of esophagus is the only tool to monitor response to treatment. Serum ultra- sensitive CRP is a non-invasive marker of inflammation in cardiovascular and gastrointestinal disorders. This study proposes to investigate the correlation of disease activity with this potential marker of inflammation in adult patients with EoE which has not been previously studied.

Specific Aim #1: To measure the baseline level of a proposed panel of inflammatory markers: serum ultra-sensitive CRP and peripheral eosinophils, as well as tissue eosinophils, mast cells, CD4 cells, IL-4, IL-5, IL-13, GM-CSF and TGF-beta in the esophagus in adult patients with eosinophilic esophagitis.

Specific Aim #2: To determine the impact of 8 week course of treatment with swallowed beclomethasone on the levels of the inflammatory markers measured in Specific Aim #1.

Specific Aim #3: To determine the correlation between the levels of the proposed panel of inflammatory markers and symptoms of EoE before and after 8 weeks of treatment with swallowed beclomethasone.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 years of age or older with biopsy proven diagnosis of EoE.
* Subjects who are able and willing to provide consent for repeat EGDs with esophageal biopsies, and blood work as per study protocol.

Exclusion criteria:

* Subjects with suspected or proven inflammatory bowel disease, malignancy, and collagen-vascular disease.
* Subjects who have used oral, inhaled or swallowed corticosteroids in the past 3 months.
* Subjects who are pregnant or breastfeeding
* Subjects who are not able to swallow beclomethasone or are intolerant to the medication.
* Subjects with history of ischemic heart disease, diabetes and dyslipidemia unless they have been stable in the last six months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Symptom improvement | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: GISOO GHAFFARI, MD, Principal Investigator — Penn State College of Medicine Hershey Medical Center
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States